CLINICAL TRIAL: NCT04468295
Title: Evaluation of the Rate of Maxillary En-masse Retraction Using 0.018-inch Versus 0.022-inch Slot Brackets in Adult Patients With Maxillary Dentoalveolar Protrusion: A Randomized Clinical Trial
Brief Title: Evaluation of the Rate of Maxillary En-masse Retraction Using 0.018-inch Versus 0.022-inch Slot Brackets in Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Abdelaziz, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBC-CU-2020-07-09
Record Dates: First submitted 2020-07-09; First posted 2020-07-13 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Orthodontic Tooth Movement
MeSH Terms: interventions — Weights and Measures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.018-inch slot orthodontic bracket system (Experimental): En-masse retraction using frictionless mechanics with 0.018-inch slot orthodontic bracket system.
  Interventions: Procedure: Bonding; Procedure: Leveling and alignment; Procedure: Extraction; Procedure: Retraction; Procedure: Digital models; Procedure: measurement
- 0.022-inch slot orthodontic bracket system (Active Comparator): En-masse retraction using frictionless mechanics with 0.022-inch slot orthodontic bracket system.
  Interventions: Procedure: Bonding; Procedure: Leveling and alignment; Procedure: Extraction; Procedure: Retraction; Procedure: Digital models; Procedure: measurement

INTERVENTIONS:
Procedure: Bonding — Bonding of upper and lower arches including 2nd maxillary molars with bracket prescription Roth 0.018 inch
Procedure: Leveling and alignment — Leveling and alignment till 0.016 x0.022 Ni Ti
Procedure: Extraction — Extraction of maxillary 1st premolars
Procedure: Retraction — En-masse retraction using 0.017x0.025 TMA T loop
Procedure: Digital models — impression taking and digital scanning
Procedure: measurement — Assessment the rate of retraction for 6 months

SUMMARY:
The study compares the rate of en-masse retraction using 0.018-inch versus 0.022-inch slot orthodontic bracket systems in adult patients with maxillary dentoalveolar protrusion.

DETAILED DESCRIPTION:
* Proper examination of the oral structures is needed to identify caries, fracture or missing teeth.
* Full set of records ( study models, lateral cephalometric radiographs, photos) will be taken for every patient as part of the routine procedure for treatment of patients in the outpatient clinic of the Orthodontic Department, Cairo University.
* In intervention group: Bonding of upper and lower arches including 2nd maxillary molars with bracket prescription Roth 0.018-inch (American Orthodontics).
* In comparator group: Bonding of upper and lower arches including 2nd maxillary molars with bracket prescription Roth 0.022-inch (American Orthodontics).
* Levelling and alignment in both groups with wire sequence: Ni-Ti (0.014,0.016, 0.016×0.022)
* Steel ligation of maxillary (2nd premolar, 1st molar and 2nd molar) for anchorage.
* Extraction of maxillary 1st premolars.
* Impression will be taken, poured in plaster from which digital models will be fabricated before beginning of en-masse retraction (the baseline model).
* Lateral cephalometric and periapical radiographs will be taken before starting retraction.
* En-masse retraction will be done using 0.017x0.025 TMA T-Loop10 in both groups, the loops will be reactivated monthly.
* Alginate impressions will be taken every month, that will be scanned to obtain digital models to assess the rate of retraction for 6 months.
* After 6 months, last obtained digital model will be evaluated for assessment of anchorage loss, and Lateral cephalometric and periapical radiographs will be taken to assess changes in the anterior teeth inclinations and apical root resorption respectively.
* The patients' treatment will be completed as indicated for them.

ELIGIBILITY:
Inclusion Criteria:

* Maxillary dentoalveolar protrusion cases that require upper first premolars extraction.
* Full permanent dentition (not necessitating third molars).
* Good oral hygiene.

Exclusion Criteria:

* Patients having systemic diseases or on medications that would affect tooth movement.
* Active periodontal disease or obvious bone loss in maxillary arch.
* Patients with habits that are detrimental to dental occlusion (thumb sucking, tongue thrusting).
* Previous orthodontic treatment.
* Missing teeth.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2020-09-28 (Estimated); Primary Completion 2021-09-28 (Estimated); Study Completion 2022-03-28 (Estimated)

PRIMARY OUTCOMES:
Retraction Rate | 6 months
  The rate of en-masse retraction of the anterior teeth

IPD SHARING:
Plan to Share IPD: No